CLINICAL TRIAL: NCT01589705
Title: Endothelial Dysfunction in Patients With Polycystic Kidney Disease
Brief Title: The Relation Between Uric Acid Level and Endothelial Dysfunction in Patients With Polycystic Kidney Disease
Status: Terminated | Type: Observational
Why Stopped: Patients recruitment and analysis were terminated
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ismail Kocyigit, TC Erciyes University Medical School, TC Erciyes University
Other Study IDs: Erciyes 2011/273
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: Uric acid; polycystic kidney disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Polycystic Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- polycystic kidney ,no hypertension: The study evaluated the association of serum uric acid levels with endothelial dysfunction in early ADPKD patients with normal renal function

SUMMARY:
There are substantial data demonstrating increased endothelial dysfunction, inflammation and oxidative stress in patients with Autosomal dominant polycystic kidney disease (ADPKD), the association between serum uric acid level and endothelial dysfunction has not been elucidated yet in these patients. Therefore, in this study, the investigators aimed to examine the relationship between the uric acid level and the ED in normotensive ADPKD patients with preserved renal function.

DETAILED DESCRIPTION:
This is the first study to evaluate the relationship between uric acid and endothelial dysfunction in patients with early stage ADPKD

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients with normal renal function,
* Normotensive ADPKD patients

Exclusion Criteria:

* Patients with impaired kidney function,
* Atherosclerotic disorders,
* Diagnosis of hypertension, gout, diabetes,
* Using of insulin, thiazide, allopurinol or uricosuric drugs

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with early stage(preserved renal function) Autosomal dominant polycystic kidney disease (n = 91) from two academic medical center.We also excluded the patients with a previous diagnosis of hypertension, gout, diabetes, current use of oral antidiabetic medication, insulin, thiazide, allopurinol or uricosuric, or a fasting glucose level 126 mg/dl. In addition, the subjects with a history of smoking or current use of any anti-hypertensive medication and statins were excluded
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Measurement of asymmetric dimethylarginine (ADMA) and flow mediated dilatation (FMD) | 4 months
  ADMA,FMD and uric acid measurements were performed to determine endothelial dysfunction in ADPKD patients

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Tokgoz, Professor, Study Director — Erciyes University Medical School
Locations (1):
- Erciyes University Medical School, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Kocyigit I, Yilmaz MI, Orscelik O, Sipahioglu MH, Unal A, Eroglu E, Kalay N, Tokgoz B, Axelsson J, Oymak O. Serum uric acid levels and endothelial dysfunction in patients with autosomal dominant polycystic kidney disease. Nephron Clin Pract. 2013;123(3-4):157-64. doi: 10.1159/000353730. Epub 2013 Jul 25. PMID 23887359